CLINICAL TRIAL: NCT00695019
Title: A Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Low-Dose Human Interferon-alpha During the 6-Month Follow-up Period of Standard Combination Therapy for Hepatitis C Virus Infection
Brief Title: Interferon-alpha Lozenges for Prevention of Relapse in Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Collaborators: CytoPharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07HWHC09
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2013-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Prevention of Relapse; HCV genotype 1b; Recurrence
MeSH Terms: conditions — Hepatitis C, Chronic; Recurrence | interventions — Interferon-alpha; Interferons

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 500 IU qd (Experimental): 500 IU Interferon-alpha lozenge taken once per day plus 2 placebo lozenges per day
  Interventions: Drug: interferon-alpha lozenges
- 500 IU tid (Experimental): 500 IU interferon-alpha lozenge taken 3 times per day
  Interventions: Drug: interferon-alpha lozenges
- placebo (Placebo Comparator): placebo lozenges taken 3 times per day
  Interventions: Drug: placebo lozenges

INTERVENTIONS:
Drug: interferon-alpha lozenges — 500 IU lozenges of natural human interferon-alpha for oral dissolution given once or three times per day for 24 weeks
  Other Names: IFN-alpha; Veldona lozenges; oral interferon; IFN-alpha lozenges; oral interferon lozenges
  Arms: 500 IU qd; 500 IU tid
Drug: placebo lozenges — 200 mg matching placebo lozenges
  Other Names: sugar pills
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether lozenges of interferon-alpha that are dissolved in the mouth can prevent relapse in patients with hepatitis C virus infection who had a complete virologic response after receiving a combination of injected interferon-alpha and oral ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* HCV genotype 1b
* Will be completing pegylated IFN-alpha and ribavirin therapy within 4 weeks
* Serum HCV RNA negative within 4 weeks of study entry

Exclusion Criteria:

* Child-Pugh score of B or C
* Decompensated liver function
* History of malignancy within past 5 years
* Other causes of liver disease besides HCV infection
* Uncontrolled diabetes or hypertension
* Unwilling to use two forms of birth control during study treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Taiwan (9):
  - Dalin Buddhist Tzu Chi General Hospital, Dalin, Chiayi County
  - Kaohsiung Chang Gung Memorial Hospital, Niaosong, Kaosiung County
  - Show-Chwan Memorial Hospital, Changhua
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Chiayi Christian Hospital, Chiayi City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - China Medical University Hospital, Taichung
  - Chang Gung Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Lee CM, Chen CY, Chien RN, Tseng KC, Peng CY, Tung SY, Fang YJ, Huang YH, Lu SN, Hung CH, Tsai TJ, Fang CC, Hsu CW, Yeh CT. A double-blind randomized controlled study to evaluate the efficacy of low-dose oral interferon-alpha in preventing hepatitis C relapse. J Interferon Cytokine Res. 2014 Mar;34(3):187-94. doi: 10.1089/jir.2013.0074. Epub 2013 Nov 15. PMID 24237300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects undergoing treatment for HCV infection at one of the 9 participating hospitals were approached, and those willing to sign informed consent were screened for eligibility.
Pre-assignment Details: A total of 196 subjects were screened. All 169 subjects meeting eligibility criteria were randomized to one of the 3 treatment groups and all 169 were included in the intent-to-treat analysis.
Groups:
- 500 IU qd: 500 IU Interferon-alpha lozenge taken once per day plus 2 placebo lozenges
Period: Overall Study
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Started | 59 | 53 | 57
Completed | 46 | 39 | 47
Not Completed | 13 | 14 | 10
Not completed — Withdrawal by Subject | 8 | 6 | 4
Not completed — Protocol Violation | 1 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Various | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 500 IU qd | 500 IU Tid | Placebo | Total
Number analyzed (Participants) | 59 | 53 | 57 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 44 | 47 | 138
  >=65 years | 12 | 9 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.9) | 55.7 (10.8) | 56.8 (9.5) | 55.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 25 | 78
  Male | 32 | 27 | 32 | 91
Region of Enrollment [Number; unit: participants]
  Taiwan | 59 | 53 | 57 | 169

OUTCOME MEASURES:

1. Secondary Outcome: Sustained Virologic Response Rate
Description: Percentage of participants who remained HCV RNA negative throughout the study
Time Frame: 48 weeks
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
percentage of participants | 71.2 | 62.3 | 66.7
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.61, Chi-squared

2. Secondary Outcome: Normalization of ALT
Description: Percentage of participants with a normal serum ALT level at the end of the study
Time Frame: 48 weeks
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
percentage of participants | 71.2 | 60.4 | 64.9
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.48, Chi-squared

3. Secondary Outcome: Change in Serum HCV RNA Concentration
Description: Change in serum HCV RNA concentration (log10 IU) from baseline to week 48
Time Frame: 48 weeks
Population: Intent-to-treat population
Measure: Log Mean (Standard Deviation); unit: log10 IU
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
log10 IU | 1.6 (2.4) | 1.9 (2.5) | 1.7 (2.5)
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.77, Kruskal-Wallis

4. Secondary Outcome: Change in Serum ALT
Description: Change in Serum ALT concentration from baseline to week 48
Time Frame: 48 weeks
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
U/L | 7.8 (75.5) | 0.6 (36.6) | 8.6 (52.6)
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.30, Kruskal-Wallis

5. Primary Outcome: Relapse Rate
Description: Percentage of participants with a positive seum HCV RNA level at any post-baseline evaluation
  Serum HCV RNA was tested using a commercially available real-time polymerase-chain-reaction (PCR) assay kit (Roche Cobas TaqMan HCV assay kit) with a limit of detection of 15 IU/ml.
Time Frame: 48 weeks
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
percentage of participants | 30.5 | 37.7 | 35.1
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.72, Chi-squared

6. Secondary Outcome: Change in Social Functioning
Description: Change in the Social Functioning domain of the SF-36 quality-of-life questionnaire from baseline to week 48
  Social Functioning (SF) scores range from 0-100, with lower scores indicating that health/emotional problems have had a greater negative impact on social activities, compared to higher scores. SF scores are calculated using a proprietary algorithm based on responses to questions #6 and #10 on the SF-36, which are 5-point likert scales about the extent to which, and the amount of time with which physical or emotional problems have interfered with social activities.
Time Frame: 48 weeks
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
change in score | 21.6 (17.7) | 16.3 (20.9) | 8.8 (20.5)
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.0023, Kruskal-Wallis — Analysis not adjusted to account for baseline differences between the groups

7. Secondary Outcome: Change in Fibrotest Score
Description: Change in fibrotest score from baseline to week 48
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 59 | 53 | 57
units on a scale | -0.37 (0.48) | -0.19 (0.46) | -0.31 (0.37)
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Fibrotest provides an estimate of liver fibrosis based on the values of 5 serum markers. Scores range from 0 to 1 with higher scores indicating a greater level of liver fibrosis. A negative change in Fibrotest score is therefore deemed to indicate improvement (reduction in fibrosis), while a positive change indicates worsening condition; Test type: Superiority or Other; p = 0.21, Kruskal-Wallis

8. Post Hoc Outcome: Normalization of Platelets
Description: Percentage of participants with a low platelet count at baseline who had a normal platelet count at the end of the study
Time Frame: 48 weeks
Population: Participants with a baseline platelet count below 150 who were evaluable for response at week 48 were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Number analyzed (Participants) | 21 | 24 | 31
percentage of participants | 81.0 | 50.0 | 41.9
Statistical Analysis 1: Comparison: 500 IU qd vs 500 IU Tid vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared
Statistical Analysis 2: Comparison: 500 IU qd vs Placebo; Test type: Superiority or Other; p = 0.005, Chi-squared

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | 500 IU qd | 500 IU Tid | Placebo
Serious Adverse Events (participants affected / at risk) | 2/59 | 6/53 | 6/57
Other Adverse Events (participants affected / at risk) | 52/59 | 46/53 | 41/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 IU qd (N=59) | 500 IU Tid (N=53) | Placebo (N=57)
Fever and loss of consciousness (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Esophageal ulcers with bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Cirrhotic liver nodule (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening of benign prostate hyperplasia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcers and anemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
right knee arthritis with synovitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Right middle cerebral artery infarction (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thoracic aortic aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness with associated nausea and vomiting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 IU qd (N=59) | 500 IU Tid (N=53) | Placebo (N=57)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6) | 7 (8)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (11) | 4 (4)
Insomnia (Nervous system disorders) | 6 (6) | 6 (6) | 6 (8)
Headache (Nervous system disorders) | 5 (7) | 4 (4) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5) | 2 (3)
Abdominal Distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Bile Duct Stone (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Malaise (General disorders) | 1 (1) | 2 (2) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No